CLINICAL TRIAL: NCT00782444
Title: Computer Navigation vs Conventional Technique in Knee Arthroplasty. A Prospective, Randomised, Clinical and Radiostereometric Trial
Brief Title: Computer Navigation vs Conventional Technique in Knee Arthroplasty
Acronym: CAOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2007/12587
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2023-01

CONDITIONS: Knee Osteoarthritis; Rheumatoid Arthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Computer navigated knee replacement (Active Comparator): Computer navigation system from Brainlab, vector vision, kolibri.
  Interventions: Procedure: Computer navigated knee replacement
- Conventional knee replacement (Placebo Comparator): Conventional total knee replacement is performed with intramedullary guides in the traditional way.
  Interventions: Procedure: Conventional knee replacement

INTERVENTIONS:
Procedure: Computer navigated knee replacement — Total knee replacement performed with the use of navigation system from Brainlab with the Profix total knee implant.
  Arms: Computer navigated knee replacement
Procedure: Conventional knee replacement — Conventional total knee replacement performed in a traditional way with the use of intramedullary rods, with the Profix implant.
  Arms: Conventional knee replacement

SUMMARY:
Project summary:

Background: Computer navigation in knee replacement surgery is increasingly being used around the world, but the documentation of its usefulness is lacking. In order to critically evaluate this new surgical method, we want to perform a prospective, randomised clinical trial.

Goal: We evaluate the need for these highly advanced techniques in knee replacement surgery, and the cost-effectiveness. Long term outcome for the patients will be predicted by using the radiostereometric analysis (RSA). Also, data from the Norwegian arthroplasty register will indicate any difference in long term survival of the implant. If there are any differences in the functional outcome or complication rate, between the two groups, this will be detected in this trial.

Method: Patients age 50 through 85 years old, with gonarthritis, in need of knee replacement, are included in the trial. Radiostereometric analysis (RSA), CT-scans, X-rays, clinical evaluation score systems and laboratory measures are used in the evaluation process. A cost-effective analysis is performed based on data from Norwegian life tables, data from SINTEF and from the Norwegian arthroplasty register. Data from the Norwegian arthroplasty register will be statistically analysed separately for all knee replacements done with computer navigation in Norway in the last 5 years. Four Norwegian hospitals will collaborate in this trial (Haukeland university hospital, Haugesund hospital, Haugesund sanitetsforenings hospital for rheumatic diseases and Lovisenberg diakonale hospital) and patients are recruited from all four hospitals.

Scientific impact/challenges: This trial will probably have great impact since good evidence supporting the use of computer navigation in knee surgery is lacking. It is important for the patient to be confident that he/she receives the best treatment, and it is important for the health care providers and funding authorities to have clear evidence when choosing between two different treatment techniques, in order for the patient to benefit.

DETAILED DESCRIPTION:
Protocol

1. Introduction: We will perform a prospective, randomized, clinically controlled RSA trial comparing:

   1. Profix cemented bicompartmental knee prosthesis implanted with conventional intramedullary instruments vs
   2. Profix cemented bicompartmental knee prosthesis implanted with the use of computer navigation (from Brainlab)

   The trial will take place at the orthopaedic departments in four hospitals: Haukeland university hospital, Haugesund hospital, Haugesund sanitetsforening rheumatism hospital and Lovisenberg diakonale hospital.The aim is to compare the technical results (implant positioning and stability) for the Profix knee prosthesis, the perioperative morbidity and the clinical and functional results comparing the two strategies. We will also evaluate the health economical aspect through a cost-effectiveness analysis. To complete the project we will analyze data from the Norwegian arthroplasty register with respect to the two different strategies. A doctoral fellowship is part of the project.
2. Background:

   In arthroplastic surgery, scientific evidence is often lacking. Haukeland university hospital in Bergen and the Norwegian arthroplasty register are closely tied, and it is natural for us to critically evaluate the usefulness and evidence of new implants and instrumentation. Computer assisted surgery is well documented in neurosurgery, but there have been a few trials in knee replacement surgery suggesting its usefulness. Some of these trials show a better alignment and positioning of the implants (1,10,12). In addition, retrospective trials have shown that the alignment is predictive of implant survival i.e. good alignment gives a better implant survival. (7,8,9) Indirectly that may indicate computer navigation is superior in regard to implant survival. Further one might assume that a better alignment gives a better functional outcome, and this new surgical technique may be less invasive, thus leading to a faster recovery. These questions still remain unanswered.
3. Challenges:

   To date there are no long term studies confirming a definite association between computer navigation and better long term results for knee replacements. No trials have thoroughly investigated the possible change in functional outcome and morbidity after the introduction of computer navigation.
4. Objectives:

We seek to find the best treatment for the osteoarthritic patients in need of a knee replacement.

1. In this trial we investigate whether there is a definite correlation between computer navigated knee replacements and a better long term survival of the implants. Radiostereometric analysis (RSA) will reveal micromotion of the implants and from other trials we know this can predict the long term survival of the implants (19,20).
2. Some trials have reported a higher perioperative morbidity for patients treated conventionally, as opposed to those treated with the assistance of computer navigation (1,11). Intramedullary rods may increase bleeding, and may give a higher frequency of postoperative delirium from microemboli and metabolic disturbances (16). On the other hand, the computer navigation is often more time consuming, and can lead to a higher risk of infection. The fixation of pin-fixators in femur and tibia for the reflection beads might weaken the bone and induce a fracture risk zone. We see that both positive and negative aspects of the computer navigation technique will be revealed in this trial.
3. The computer navigation software, hardware and surgical instruments add costs to the knee replacement procedure. Hence, it is important to evaluate the benefit as compared to the costs. We will analyze this using registry data and a Markov decision analysis.
4. The Norwegian arthroplasty register has data from all Norwegian hospitals. These data will be analyzed and published with regard to computer navigated knee replacement.

5) Method: We will randomize Profix cemented bicompartmental total knee implanted conventionally vs the same prosthesis implanted with the assistance of computer navigation. Profix is the standard implant in Helse Vest and it has good 5-year implant survival data in our Norwegian arthroplasty register (15).Tantalum markers will be injected into the bone and the implant for radiostereometric analysis (RSA). The radiographic technique is somewhat challenging and we have recruited specially trained and educated radiographers to obtain these images.The images allow us to localize every marker in a three dimensional coordinate system. Mathematic models will then calculate differences in position from one image to another. Micromotion down to 0,1mm and 0,2 degrees will be detected. Micromotions within the first two years correlate with long term implant survival. The radiation dose is low (10-20% of a regular x-ray of the knee). The image processing and the calculations are time consuming and expensive. Special software is needed and we therefore collaborate with Kompetansesenter for ortopediske implantater by Norges teknisk-naturvitenskapelige universitet (NTNU).

Prior to the inclusion of patients, every surgeon has performed more than 10 knee replacements with computer assistance. All surgeons are skilled and have performed more than 100 knee replacements with the conventional technique. A pilot study with 12 patients (6 in each group) will be performed. A total of 200 patients (100 in each group) will be included in the trial.

Only 60 patients will be included in the RSA part of the trial. The precision of the RSA will be evaluated by double investigations at a 1-year follow-up. The patient receives two images separated by a short period of time. The patient is first radiographed, then he/she takes a walk in the investigation room, and is then radiographed again. Micromotion between these two images is not real, so then we know the precision of our method. The limits for significant differences are calculated as 99% confidence intervals of absolute differences for the double investigation. The upper limits for "mean error of rigid body fitting" and "condition number" are set to 0,35mm and 130. These parameters describe the stability of the marker and the spreading, and expresses the precision of the software. At least 20 patients are needed in each group, but the technical demanding procedure has a drop-out risk, leading us to include 30 patients in each group (23).

We aim to reveal a difference of 0,5 degrees in the two groups with alignment in the frontal plane as measured on the CT-scan. Earlier research in this field indicates a greater variation in the conventional group (standard deviation=1,3) than in the computer navigated group (standard deviation=0,9) (10). With 80% statistical power and a significance level of 0.05, a power calculation suggests 79 patients in each group. Further, to be able to detect a difference of 10 units in our functional score (KOOS)(13) with a common standard deviation of 20 (14), our power calculations suggested 94 patients in each group to reach a power of 80% at a significance level of 0,05. From these calculations we chose a study design with 100 patients in each group, assuming there will be some drop-outs. The study is recommended by the Regional ethics committee, Personvernombudet for forskning (Norsk samfunnsvitenskapelig datatjeneste) and Statens strålevern.

In the 10-years follow-up, the following analyses will be performed (two publications are planned):

Publication 1 - Pain Trajectories After TKA

Aims:

To identify latent classes of patients based on their pain trajectories (measured by KOOS Pain) over a 10-year period following total knee arthroplasty (TKA).

To evaluate factors associated with class membership, including:

Sociodemographic variables Disease status and comorbidities Clinical factors (e.g., surgical time, radiological findings, CAS vs conventional technique) EQ-5D Anxiety/Depression EQ VAS (self-reported health status)

Statistical Analysis:

Latent Class Analysis (LCA) or Growth Mixture Modeling (GMM) for trajectory identification.

Logistic or multinomial regression to assess associated factors (depending on the number of classes).

Publication 2 - ADL/Function After TKA

Aims:

To identify latent classes of patients based on their knee-specific function/ADL scores (measured by KOOS ADL) over a 10-year period following TKA.

To evaluate factors associated with class membership, including:

Sociodemographic variables Disease status and comorbidities Clinical factors (e.g., surgical time, radiological findings, CAS vs conventional technique) EQ-5D Anxiety/Depression EQ VAS (self-reported health status)

Statistical Analysis:

Latent Class Analysis (LCA) or Growth Mixture Modeling (GMM) for trajectory identification.

Logistic or multinomial regression to assess associated factors (depending on the number of classes).

6) Main activities and milestones: Cost-effectiveness analysis 2010 Inclusion and surgery, 2010 Analyzing CT scans and functional results, spring and summer 2012 Publication of 3 months follow-up, fall 2012 Analyzing RSA results 2012/2013 Publication of RSA results 2012/2013 Register analysis, 2010/2012 PROMS analysis including investigation of trajectories of pain and function for the two methods 2025 (10-years-follow-up-data)

7)Scientific impact: There are many new and expensive instrumentations and implants on the market today. In order for Norwegian hospitals to be able to offer a high international standard of treatment, we need to evaluate carefully before choices are made. To date, computer navigation in knee replacement surgery is not well documented to be recommended as a standard procedure at all Norwegian hospitals. Earlier studies are lacking in that they have not reported an impact on long term implant survival. This study is unique by using RSA to predict long term outcome. It is also large enough to evaluate functional results and morbidity. In addition, the register analysis will give us information that has not been published. It is important for the patient to be confident that he/she receives the best treatment available, and it is important for the health care providers and funding authorities to receive clear and accurate information when choosing between two different treatments, in order to gain the most benefit.

8)Dissemination of project results: We will publish our results in high impact international medical journals to disseminate the results to colleagues around the world. Lectures and presentations in national and international congresses is a natural way to publish the results. An investigator education programme, PhD, is incorporated in the project, which includes presentations and posters in national and international congresses. The project will be registered in an international trial register, according to demands by many journals before publishing.

ELIGIBILITY:
Inclusion Criteria:

* men and women age 50-85 years old
* primary and secondary knee osteoarthritis
* rheumatic arthritis of the knee
* well compensated heart or lung disease(ASA-grad 1-3)
* patients recruited from orthopaedic departments at Haugesund hospital og Haugesund Sanitetsforenings Revmatismesjukehus, Haukeland university hospital, Lovisenberg Diakonale hospital
* informed consent
* MMS-score > 20 elir. , tas MMS også dag 2
* Hb > 11,5 for women and Hb > 13 for men

Exclusion Criteria:

* advanced systemic disease
* general or local infection
* neurological or myogenic disease
* Paget's disease of bone
* bone cysts in the tibia or femur > 2 cm in diameter and within 2 cm from the articular surface
* liver disease
* uncontrolled haematological disease
* B-TRC < 165
* B-Hb < 11,5 for women
* B-Hb < 13 for men
* cancer
* uncontrollable heart or lung disease (ASA-class 4)
* dementia
* immobile hips
* hip replacement in ipsilateral hip
* knee injury < 1år earlier
* metal allergy
* extreme valgus deformity > 15 degrees or curvature of the tibia, necessitating extramedullary device
* earlier fracture of the femur makes it impossible to use intramedullary rod Osteotomy of the proximal tibia og distal femur
* BMI > 35
* Only one knee recruited per patient

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2009-01; Primary Completion 2023-01 (Actual); Study Completion 2023-01 (Actual)

PRIMARY OUTCOMES:
longevity of the implant | 2yrs for RSA, 10 yrs in vivo

SECONDARY OUTCOMES:
Function of the knee | 2 yrs
Bleeding | 1 week
complications | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ove Furnes, Phd, MD, Study Director — Haukeland University Hospital
Locations (4):
- Norway (4):
  - Haugesund sanitetsforenings revmatismesykehus, Haugesund, Haugesund
  - Lovisenberg diakonale sykehus, Oslo, Oslo County
  - Haukeland university hospital, Bergen
  - Haugesund hospital, Haugesund

REFERENCES:
- [Background] Chauhan SK, Scott RG, Breidahl W, Beaver RJ. Computer-assisted knee arthroplasty versus a conventional jig-based technique. A randomised, prospective trial. J Bone Joint Surg Br. 2004 Apr;86(3):372-7. doi: 10.1302/0301-620x.86b3.14643. PMID 15125124
- [Background] Luring C, Bathis H, Tingart M, Perlick L, Grifka J. Computer assistance in total knee replacement - a critical assessment of current health care technology. Comput Aided Surg. 2006 Mar;11(2):77-80. doi: 10.3109/10929080600578925. PMID 16782642
- [Background] Chauhan SK, Clark GW, Lloyd S, Scott RG, Breidahl W, Sikorski JM. Computer-assisted total knee replacement. A controlled cadaver study using a multi-parameter quantitative CT assessment of alignment (the Perth CT Protocol). J Bone Joint Surg Br. 2004 Aug;86(6):818-23. doi: 10.1302/0301-620x.86b6.15456. PMID 15330021
- [Background] Furnes O, Espehaug B, Lie SA, Vollset SE, Engesaeter LB, Havelin LI. Failure mechanisms after unicompartmental and tricompartmental primary knee replacement with cement. J Bone Joint Surg Am. 2007 Mar;89(3):519-25. doi: 10.2106/JBJS.F.00210. PMID 17332100
- [Background] Rand JA, Coventry MB. Ten-year evaluation of geometric total knee arthroplasty. Clin Orthop Relat Res. 1988 Jul;(232):168-73. PMID 3383484
- [Background] Ritter MA, Faris PM, Keating EM, Meding JB. Postoperative alignment of total knee replacement. Its effect on survival. Clin Orthop Relat Res. 1994 Feb;(299):153-6. PMID 8119010
- [Background] Fehring TK, Odum S, Griffin WL, Mason JB, Nadaud M. Early failures in total knee arthroplasty. Clin Orthop Relat Res. 2001 Nov;(392):315-8. doi: 10.1097/00003086-200111000-00041. PMID 11716402
- [Background] Bathis H, Shafizadeh S, Paffrath T, Simanski C, Grifka J, Luring C. [Are computer assisted total knee replacements more accurately placed? A meta-analysis of comparative studies]. Orthopade. 2006 Oct;35(10):1056-65. doi: 10.1007/s00132-006-1001-3. German. PMID 16953328
- [Background] Roos EM, Toksvig-Larsen S. Knee injury and Osteoarthritis Outcome Score (KOOS) - validation and comparison to the WOMAC in total knee replacement. Health Qual Life Outcomes. 2003 May 25;1:17. doi: 10.1186/1477-7525-1-17. PMID 12801417
- [Background] Hallan G, Aamodt A, Furnes O, Skredderstuen A, Haugan K, Havelin LI. Palamed G compared with Palacos R with gentamicin in Charnley total hip replacement. A randomised, radiostereometric study of 60 HIPS. J Bone Joint Surg Br. 2006 Sep;88(9):1143-8. doi: 10.1302/0301-620X.88B9.18008. PMID 16943462
- [Background] Ryd L, Albrektsson BE, Carlsson L, Dansgard F, Herberts P, Lindstrand A, Regner L, Toksvig-Larsen S. Roentgen stereophotogrammetric analysis as a predictor of mechanical loosening of knee prostheses. J Bone Joint Surg Br. 1995 May;77(3):377-83. PMID 7744919
- [Derived] Gothesen O, Espehaug B, Havelin LI, Petursson G, Hallan G, Strom E, Dyrhovden G, Furnes O. Functional outcome and alignment in computer-assisted and conventionally operated total knee replacements: a multicentre parallel-group randomised controlled trial. Bone Joint J. 2014 May;96-B(5):609-18. doi: 10.1302/0301-620X.96B5.32516. PMID 24788494